CLINICAL TRIAL: NCT04863560
Title: Brain Activity Response to Cues During Gait in Parkinson's
Brief Title: Brain Activity During Gait in Parkinson's
Acronym: BARC-PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Collaborators: Parkinson's Foundation (Other); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PF-CRA-2073; 286383 (Other: IRAS); 20/LO/1036 (Other: NHS Research Ethics Committee Reference)
Record Dates: First submitted 2021-04-06; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
Keywords: Parkison's disease; Gait; functional near infrared spectroscopy; electroencephalography; Inertial Sensors; Brain activity; Cueing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hoehn & Yahr stage I (H&YI): - 20 Hoehn & Yahr stage I (early disease, minimal symptoms)
  Interventions: Other: Auditory Cueing; Other: Visual Cueing; Other: tactile Cueing
- Hoehn & Yahr stage II (H&YII): - 30 Hoehn & Yahr stage II (mild disease, no balance issues)
  Interventions: Other: Auditory Cueing; Other: Visual Cueing; Other: tactile Cueing
- Hoehn & Yahr stage III (H&YIII): - 30 Hoehn & Yahr stage III (moderate disease, balance issues)
  Interventions: Other: Auditory Cueing; Other: Visual Cueing; Other: tactile Cueing

INTERVENTIONS:
Other: Auditory Cueing — Metronome beat to step in time with
Other: Visual Cueing — Lines on the floor to step over
Other: tactile Cueing — Vibration to step in time with (metronome like)

SUMMARY:
Lay Summary:

Walking problems, such as slow and short steps, are very common in Parkinson's disease and lead to increased falls risk, as well as reduced mobility and quality of life. Walking issues are difficult to treat as medication interventions do not restore walking ability in people with Parkinson's, therefore physiotherapy approaches are used to help improve walking. Various physiotherapy strategies have been used, such as internal (thinking about bigger steps) or external prompts. External prompts include auditory (a metronome beat to step in time to), visual (lines to step over on the floor) and tactile (metronome-like vibration to step with) prompts that are very commonly used to improve walking in Parkinson's. However, the reason why walking improves in people with Parkinson's with these physiotherapy strategies is unknown, which has led to not all patients benefiting and only short-term walking improvements being seen.

The main issues are that it is unclear if these various internal or external prompt strategies are effective with the progression of Parkinson's disease, and it is unknown which type of strategy is most effective at different disease stages or with more severe walking impairment, such as freezing (the inability to progress walking for short periods despite wanting to do so). Being able to use specific brain regions to pay attention to different internal or external prompts has been suggested to be the reason why people with Parkinson's can overcome their walking problems, but this has not been tested. Therefore, this study will use state-of-the-art digital technology to measure walking and brain activity changes with different internal and external prompts. The investigators think that the walking improvement with different prompt strategies relies on the ability to activate specific brain regions, and that brain region activity in response to internal or external prompts will change at different stages of Parkinson's disease.

Ultimately, understanding the reasons why people benefit from these physiotherapy strategies and who benefits most from specific strategies will enable clinicians to provide more timely and efficient treatment for people with Parkinson's, and to develop more effective strategies to further improve walking.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's by a movement disorder specialist according to United Kingdom (UK) brain bank criteria
* Hoehn & Yahr (H&Y) stage I-III
* Aged >50 years
* Able to walk and stand unaided
* Adequate hearing (as evaluated by the whisper test; stand 2m behind subject and whisper a 2 syllable word, subject repeats word) and vision capabilities (as measured using a Snellen chart - 6/18-6/12).
* Stable medication for the past 1 month and anticipated over a period of 6 months

Exclusion Criteria:

* Psychiatric co-morbidity (e.g., major depressive disorder as determined by Geriatric Depression Scale - short form (GDS-15); <10 [26])
* Clinical diagnosis of dementia or other severe cognitive impairment (Montreal cognitive assessment <21 [27])
* History of stroke, traumatic brain injury or other neurological disorders (other than PD, for the PD group)
* Acute lower back or lower extremity pain, peripheral neuropathy, rheumatic and orthopaedic diseases
* Unstable medical condition including cardio-vascular instability in the past 6 months
* Unable to comply with the testing protocol or currently participating in another interfering research project
* Interfering therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve 80 participants with PD, who will be split into groups dependent on the severity of their disease (classified with the Hoehn and Yahr (H&Y) scale); n=20 H&Y stage I (early disease, minimal symptoms); n=30 H&Y stage II (mild disease, no balance issues); n=30 H&Y stage III (moderate disease, balance issues).
  Within the H&Y stage II and III groups, we will also ensure recruitment of a sub-group of n=15 individuals who self-report FOG within each group (n=30 total with FOG), which will provide a sub-group for further data analysis. We will limit FOG sub-group recruitment to these groups as we do not expect any individuals with FOG to be in H&Y stage I.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in cortical oxygenated hemoglobin (HbO2) signal during walking | immediately after intervention
  Change in cortical oxygenated hemoglobin (HbO2) measured while walking with cueing, which will be quantified with a wireless functional near infrared spectroscopy (fNIRS) system
Change in cortical power spectral densities during walking | immediately after intervention
  Change in cortical power spectral densities of EEG signals from cortex with cueing, which will be quantified with a mobile electroencephalography (EEG) system

SECONDARY OUTCOMES:
Change in Stride Length (m) | immediately after intervention
  Change in stride length with cueing
Change in Gait Speed (m/s) | immediately after intervention
  Change in speed of walking with cueing
Change in Stride Time (s) | immediately after intervention
  Change in time taken to complete a stride when walking with cues
Change in Gait Variability (SD) | immediately after intervention
  Change in variability (standard deviation; SD) of gait when walking with cues

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Stuart, PhD, Principal Investigator — Northumbria University
Locations (3):
- Oregon Health & Science University, Portland, Oregon, United States
- United Kingdom (2):
  - Northumbria University, Newcastle upon Tyne
  - Northumbria Healthcar NHS foundation trust, North Shields

IPD SHARING:
Plan to Share IPD: Yes
Access to the datasets can be obtained by contacting the principle investigator.

REFERENCES:
- [Derived] Vitorio R, Morris R, Das J, Walker R, Mancini M, Stuart S. Brain activity response to cues during gait in Parkinson's disease: A study protocol. PLoS One. 2022 Nov 17;17(11):e0275894. doi: 10.1371/journal.pone.0275894. eCollection 2022. PMID 36395190
- See also: Physiotherapy Innovation Laboratory Website — http://www.pi-lab.co.uk

DOCUMENTS (1):
  • Informed Consent Form (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04863560/ICF_000.pdf